CLINICAL TRIAL: NCT04281836
Title: Visual and Auditory Neuromodulation of Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, MS, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00100981
Record Dates: First submitted 2020-02-13; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Pain, Acute
Keywords: fNIRS; Virtual Reality (VR); Breathing focusing based meditation
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing awareness through use of virtual reality breathing (Experimental): Healthy participants were recruited in this group.
  Interventions: Behavioral: Interoceptive breathing awareness through use of audio and visual virtual technology aid
- Traditional breathing awareness (Active Comparator): Healthy participants were recruited in this group.
  Interventions: Behavioral: Interoceptive breathing awareness without use of audio or visual virtual reality

INTERVENTIONS:
Behavioral: Interoceptive breathing awareness through use of audio and visual virtual technology aid — Participants are asked to focus on their breathing while (a) listening to their breathing sounds with headphones and (b) watching the 3-D image of their lungs inhaling and exhaling in real-time using the Oculus Rift 3D virtual imaging equipment and plethysmography belt. During this time fNIRS and tQST data will be collected (more detail provided below).
  Arms: Breathing awareness through use of virtual reality breathing
Behavioral: Interoceptive breathing awareness without use of audio or visual virtual reality — Participants are asked to focus on their breathing. During this time fNIRS and tQST data will be collected (more detail provided below).
  Arms: Traditional breathing awareness

SUMMARY:
Medical and dental patients may experience fear commonly attributed to physical pain during the visit. By reducing pain perception, patient comfort and future patient compliance may be improved. Patient health may be improved by increasing compliance and promoting increased visits. This can lead to more frequent and timely preventative actions. The research purpose is to establish quantitative and qualitative data to support current, non-pharmacological methods for reducing pain sensitivity. More specifically, the investigators aim to determine if the use of auditory and visual (3D imaging) stimuli related to the regulation of breathing can decrease or modulate pain.

Healthy participants between the ages of 18 and 60 will participate in a one week study, with two in lab appointments on day one and day seven. Participants will be split into two groups, one will undergo breathing awareness using auditory and visual technology (i.e. listen to one's own breathing with headphones and watch 3D image of lungs using virtual headset), and the second group will have breathing awareness without the use of technology (i.e. simply focusing on one's own breathing). At each appointment, the investigators will collect pain threshold data using thermal Quantitative Sensory Testing (tQST) and brain activity data using Functional near-infrared spectroscopy (fNIRS). tQST and fNIRS data will be collected before, during, and after each breathing awareness/control exercise.

Quantifying change in pain intensity has been demonstrated by pain threshold comparison across a stimulus using thermal Quantitative Sensory Testing (tQST). Functional near-infrared spectroscopy (fNIRS) in coordination with pain stimulation has been shown effective at locating different hemodynamic cortical responses depending on pain perception and expectation. In the current study, functional resting states before and after pain stimulation will be quantitatively assessed using fNIRS.

The study design will allow the investigators to determine if the use of auditory and visual (3D imaging) stimuli related to the regulation of breathing can decrease or modulate pain. Cortical responses will give additional insight into the areas related to the decreased pain threshold. The long term objective is to increase neurophysiological understanding that will improve patient care. If effective, the novel experimental methods used will help to standardize future pain evaluation techniques.

DETAILED DESCRIPTION:
The study requires seven consecutive days of participation: two in-person appointments, day 1 and 7, and at home self-guided exercises days 2-7 Both in-person appointments will be held at the fNIRS lab at the University of Michigan Center for Human Growth and Development. The participants will be randomly divided into two even groups:

1. Interoceptive breathing awareness through the use of audio and visual virtual technology aid Participants are asked to focus on their breathing while (a) listening to their breathing sounds with headphones and (b) watching the 3-D image of their lungs inhaling and exhaling in real-time using the Oculus Rift 3D virtual imaging equipment and plethysmography belt. During this time fNIRS and tQST data will be collected (more detail provided below).
2. Control: Interoceptive breathing awareness without the use of audio or visual virtual technology aid Participants are asked to focus on their breathing. During this time fNIRS and tQST data will be collected (more detail provided below).

Each in-person appointment is anticipated to last one hour, with 3x daily at-home sessions lasting 5 minutes each. Instructions for at-home sessions will be provided. Each participant is to complete all 7 sessions in 7 consecutive days plus or minus one day. The total time commitment is3hours 15 minutes. In the advent of equipment malfunction during a session that compromises or prevents data collection, the participant may be asked to return for an additional appointment to complete the session.

The first session will begin with documentation of subject consent followed by the completion of a demographic survey. At the start of all sessions, subjects will be asked to complete questionnaires on their current pain levels and emotional states, including the McGill Pain Questionnaire (MPQ) and Positive and Negative Affect Schedule (PANAS). Baseline thermal quantitative sensory testing (tQST) data will also be collected by 3 trials of heat administration (more detail provided below). Participants will then be seated in a dental chair wearing headphones, Oculus Rift 3D virtual imaging equipment, plethysmography belt , fNIRS sensors, thermal quantitative sensory (tQST) sensors with holding apparatus, and a pulse oximeter. A single, unilateral tQST sensor will be localized to the left mandibular nerve branch of the trigeminal cranial nerve, V3. The fNIRS sensors will be worn on the head and positioned for optimal brain imaging. All fNIRS data will be collected and analyzed with Homer 2 software. The pulse oximeter will be clipped over one finger to measure general body blood oxygen content during the session.

Once the participant is seated, wearing the equipment and hooked up to the fNIRS device, the following will take place for the two breathing awareness experimental sessions:

1. Participants will be asked to relax for five minutes to allow baseline data collection of the patient's resting functional state.
2. After 5 minutes of baseline collection, interoceptive breathing awareness (with or without the use of technology) will begin for a period of 10 minutes, during which fNIRS and pulse oximeter data will be collected.
3. After 10 minutes of the breathing awareness exercise, the thermal QST will begin using the Medoc (Israel) Pathway System. The holding apparatus with the QST system will administer a hot stimulus at a consistent location and pressure from a baseline temperature of 30 Celsius (86 Fahrenheit), for reference the average normal body temperature is 37 Celsius (98.6 Fahrenheit). The participant will control the heating unit with a computer keyboard. The temperature will gradually increase 1 Celsius per second up to 50 Celsius (122 Fahrenheit). At the first detection of pain, the subject will be instructed to click the keyboard space bar to stop the temperature from increasing. This process will be repeated twenty times to give an accurate average temperature value. During the 20 trials, participants will continue the interceptive breathing awareness and fNIRS and pulse oximeter data will continue to be collected.
4. Upon completion of all 20 tQST trials, participants will be asked to discontinue the breathing awareness exercise and five minutes of resting functional state will again be collected. Once resting state is collected, all equipment and sensors will be turned off and removed from the participant, at which point the participant will again complete the mood and pain surveys and 3 trials of post-stimulation tQST data will be collected.

Audio and Visual Virtual Technology: Headphones, microphone, and the Oculus Rift will be connected to the mobile device. Breathing sounds will be picked up by a microphone and played back to the participant through the headphones. The sounds of inhaling and exhaling will be identified by the app and the respiratory volume will be identified via a plethysmography belt allowing proper synchronization of the virtual lung image on the Oculus with the participant's own lungs. The processing and replay of this information will occur in less than a second allowing the participant to experience the virtual environment in real-time. (I.e. Participants will be able to see a 3D image of their lungs inflating and deflating, while at the same time listening to their breathing, for a truly immersive experience).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-60
* Healthy subjects with no ongoing medical conditions

Exclusion Criteria:

* Significant hearing and visual impairment
* Concurrent use of opioids or NSAIDs
* History or current evidence of chronic pain; recent acute pain during the past 6 months
* History of neurological disorder (e.g. epilepsy, stroke, neuropathy, neuropathic pain)
* History or current evidence of a psychotic disorder (e.g. schizophrenia) or substance abuse by Diagnostic and Statistical Manual of Mental Disorders - IV; bipolar or severe major depression
* Ongoing, unresolved disability litigation
* Use of an investigational drug or device within 30 days of study entry
* Pregnancy during course of study
* History or current evidence of respiratory distress or asthma
* History of uncontrolled endocrine disturbances (diabetes, thyroid, etc.)
* Any severe clinical condition that in the opinion of the PI interferes with the study
* Beards and/or facial hair
* Inability complete all sessions within 7 days plus or minus one day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in pain threshold | Baseline, 7 days
  Pain threshold will be measured by thermal stimulation. During the thermal stimulation, a single, unilateral thermal quantitative sensor was localized to the left mandibular nerve branch of the trigeminal cranial nerve, V3. The thermal quantitative sensory test (tQST) administered a hot stimuli at a consistent location and pressure from a baseline temperature of 30 Celsius (86 Fahrenheit), for reference the average normal body temperature is 37 Celsius (98.6 Fahrenheit ), to a maximum temperature of 50 Celsius (122 Fahrenheit). Once the trial is initiated on the computer, the temperature on the thermal sensor gradually increased 1 Celsius per second. The participant was in control the heating unit with a remote and was instructed to push the button on the remote at the first detection of pain; this stopped the temperature from increasing and recorded the pain threshold.
The Positive and Negative Affect Schedule (PANAS) Score | Baseline (day 1)
  PANAS is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). The participants were asked to fill this questionnaire to report their emotional status before and after the breathing training and thermal stimulation sessions.
The Positive and Negative Affect Schedule (PANAS) Score | Day 7
  PANAS is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). The participants were asked to fill this questionnaire to report their emotional status before and after the breathing training and thermal stimulation sessions.
Functional near-infrared spectroscopy (fNIRS) neuroimaging data | Baseline (day 1)
  fNIRS is an optical neuroimaging technique. We applied 15 light emitters and 22 light detectors, yielding 45 data recording channels. We deployed these channels at bilateral prefrontal, sensory, and visual cortices to collect neuroimaging data during resting state, breathing training, and thermal stimulation sessions.
Functional near-infrared spectroscopy (fNIRS) neuroimaging data | Day 7
  fNIRS is an optical neuroimaging technique. We applied 15 light emitters and 22 light detectors, yielding 45 data recording channels. We deployed these channels at bilateral prefrontal, sensory, and visual cortices to collect neuroimaging data during resting state, breathing training, and thermal stimulation sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre FM DaSilva, DMedSc, Principal Investigator — School of Dentistry, University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States